CLINICAL TRIAL: NCT00279214
Title: An Evaluation of Vasopressor Requirement, Hemodynamic Response and Measures of Tissue Perfusion With the Administration of Drotrecogin Alfa (Activated) as Part of Physician-Directed Therapy in Patients With Septic Shock
Brief Title: Hemodynamic and Perfusion Response to Drotrecogin Alfa (Activated) in Patients With Septic Shock
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9944; F1K-US-EVDA
Record Dates: First submitted 2005-12-15; First posted 2006-01-19 (Estimated); Results first posted 2009-08-17 (Estimated); Last update posted 2009-09-02 (Estimated); Status verified 2009-08

CONDITIONS: Sepsis; Septic Shock
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — drotrecogin alfa activated

INTERVENTIONS:
Drug: drotrecogin alfa (activated)

SUMMARY:
The study will evaluate the vasopressor requirement, hemodynamic response and measures of tissue perfusion in patients with septic shock receiving an infusion of drotrecogin alfa (activated) compared to patients not receiving drotrecogin alfa (activated).

ELIGIBILITY:
Inclusion:

* 18 years of age or older with a diagnosis of septic shock
* presence of a pulmonary artery catheter (or central venous catheters)
* requiring vasopressor support despite adequate fluid resuscitation
* an intravenous steroid administered for septic shock, except for those patients who were tested and are responders to a corticotropin stimulation test, or patients who do not receive a steroid due to the clinical judgment of the treating physician, based on an alternate assessment (e.g. normal baseline cortisol).

Exclusion:

* Onset of first-sepsis induced organ dysfunction is greater than 24 hours from the time of informed consent
* Baseline measurements of pulmonary artery occlusive pressure (PAOP) < 12 mmHg or a central venous pressure (CVP) < 8 mmHg
* Patient requires continuous oxygen therapy by face-mask
* The presence of an advanced directive to withhold life-sustaining treatment, with the exception of a directive to withhold chest compressions only
* Have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry
* Weight > 200 kg
* Are moribund (not expected to survive 24 hours)
* Are pregnant or are lactating and the milk is to be ingested by the infant (pregnancy status must be verified by urine or serum testing)
* Have not completed written informed consent signed by the patient or the patient's legal representative.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2005-11; Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-651-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Camden, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Akron, Ohio

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Although 22 and 21 patients were randomized to drotrecogin alfa (activated) [DrotA(a)] and control, respectively, 3 patients in DrotA(a) and 2 patients in control did not receive the per-protocol treatment, and as such, they have been excluded from the baseline demographics and the per-protocol efficacy analyses.
Groups:
- Drotrecogin Cohort: Group received drotrecogin alfa (activated) per physician-directed therapy
- Control Cohort: Group did not receive drotrecogin alfa (activated) per physician-directed therapy
Period: Overall Study
Arm/Group | Drotrecogin Cohort | Control Cohort
Started | 22 | 21
Completed | 19 (Completed means the number of per-protocol patients in the study) | 19 (Completed means the number of per-protocol patients in the study)
Not Completed | 3 | 2
Not completed — Physician Decision | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Drotrecogin Cohort | Control Cohort | Total
Number analyzed (Participants) | 19 | 19 | 38
Age Continuous [Mean (Standard Deviation); unit: years] | 68.0 (11.8) | 65.8 (15.0) | 66.9 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 11 | 12 | 23
Region of Enrollment [Number; unit: participants]
  United States | 19 | 19 | 38
Race/Ethnicity [Number; unit: participants]
  African | 1 | 1 | 2
  Caucasian | 16 | 15 | 31
  East Asian | 1 | 0 | 1
  Hispanic | 1 | 3 | 4
Cardiac Index [Mean (Standard Deviation); unit: liters/minute/meters squared] — Cardiac Index = cardiac output divided by body surface area.
  liters/minute/meters squared | 3.5 (1.7) | 3.3 (1.4) | 3.4 (1.6)
Creatinine Clearance [Mean (Standard Deviation); unit: milliliter per minute] — CrCl = (urine creatinine*urine volume)/(plasma creatinine*time period of urine collection). Corrected CrCl = CrCl*1.73/body surface area. Change in CrCl = Endpoint minus baseline.
  milliliter per minute | 69.2 (77.0) | 29.9 (31.1) | 52.9 (64.5)
Cumulative Vasopressor Index (CVI) [Mean (Standard Deviation); unit: units on a scale] — CVI is sum of rankings for all vasopressors being used by patient at given time.
  Based on relative potency and dosing range for each vasopressor, each vasopressor was assigned ranking of 1 (low dosage) to 4 (high dosage). Range of CVI is between
  1 and 20.
  units on a scale | 4.3 (2.1) | 4.4 (2.4) | 4.4 (2.2)
Lactate Levels [Mean (Standard Deviation); unit: millimoles per Liter] — Measures of global tissue perfusion and oxygenation were assessed via lactate levels.
  millimoles per Liter | 2.0 (1.1) | 2.6 (2.8) | 2.3 (2.1)
Mean Arterial Pressure (MAP) [Mean (Standard Deviation); unit: mm Hg] | 73.5 (9.9) | 72.1 (9.4) | 72.8 (9.5)
Mixed Venous Oxygen Saturation [Mean (Standard Deviation); unit: percent saturation mixed venous oxygen] — Cardiovascular performance measures obtained with a pulmonary catheter as assessed by mixed venous oxygen saturation.
  percent saturation mixed venous oxygen | 68.9 (15.6) | 68.9 (10.1) | 68.9 (12.9)
Number of Organ Dysfunctions [Mean (Standard Deviation); unit: number of organ dysfunctions] | 2.5 (0.8) | 2.0 (0.9) | 2.3 (0.9)
Ratio of Arterial Partial Pressure of Oxygen to Fraction of Inspired Oxygen (PaO2/FiO2) [Mean (Inter-Quartile Range); unit: mm Hg / percent inspired oxygen] | 191.8 [140.0 to 260.0] | 248.3 [181.7 to 330.0] | 222.0 [164.0 to 303.3]
Total Sequential Organ Failure Assessment Score [Mean (Standard Deviation); unit: units on a scale] — The presence of 5 organ dysfunctions (cardiovascular, respiratory, renal, hepatic, coagulation) was assessed using a Sequential Organ Failure Assessment (SOFA) score. Each organ has a possible dysfunction score of 0 to 4, for a total SOFA score range of 0 (no organ dysfunction) to 20 (all organs with dysfunction).
  units on a scale | 8.5 (2.0) [7 to 10] | 8.3 (3.2) [6 to 10] | 8.4 (2.6) [6 to 10]

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Vasopressor Index (CVI)
Description: CVI is sum of rankings for all vasopressors being used by patient at given time. Based on relative potency and dosing range for each vasopressor, each vasopressor was assigned ranking of 1 (low dosage) to 4 (high dosage). Range of CVI is between 1 and 20.
Time Frame: baseline to 24 hours
Population: Number of per-protocol participants with values at baseline and 24 hours.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Drotrecogin Cohort | Control Cohort
Number analyzed (Participants) | 19 | 19
units on a scale
  24 Hour | 2.3 (2.5) | 3.0 (2.8)
  24 Hour Change from Baseline | -2.0 (2.2) | -1.4 (2.2)
Statistical Analysis 1: Comparison: Drotrecogin Cohort vs Control Cohort; 24-Hour p-value; Test type: Superiority or Other; p = 0.238, Repeated Measures - propensity adjusted
Statistical Analysis 2: Comparison: Drotrecogin Cohort vs Control Cohort; Test type: Superiority or Other; p = 0.281, Repeated Measures - propensity adjusted — 24-Hour Change from Baseline p-value

2. Secondary Outcome: Change From Baseline to 96 Hour Endpoint in Cumulative Vasopressor Index (CVI)
Description: as for outcome 1
Time Frame: Baseline, 96 hours
Population: Number of per-protocol participants with values at baseline and 96 hours.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Drotrecogin Cohort | Control Cohort
Number analyzed (Participants) | 18 | 16
units on a scale
  96 Hour | 0.4 (1.3) | 0.5 (1.4)
  96 Hour Change from Baseline | -3.7 (2.5) | -3.3 (2.1)
Statistical Analysis 1: Comparison: Drotrecogin Cohort vs Control Cohort; Test type: Superiority or Other; p = 0.478, Mixed Models Analysis — P-value for 96 Hour Change from Baseline; Model: Outcome=Therapy + Sedative Indicator + Time + Therapy*Time + Propensity Score

3. Secondary Outcome: Mean Arterial Pressure
Time Frame: baseline to 24 hours
Population: Number of per-protocol participants with values at baseline and 24 hours.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Drotrecogin Cohort | Control Cohort
Number analyzed (Participants) | 19 | 18
mm Hg
  24 Hours | 78.2 (11.3) | 75.6 (9.8)
  24 Hour Change from Baseline | 4.7 (14.6) | 2.5 (12.4)
Statistical Analysis 1: Comparison: Drotrecogin Cohort vs Control Cohort; Test type: Superiority or Other; p = 0.442, Repeated Measures - propensity adjusted — 24-Hour p-value
Statistical Analysis 2: Comparison: Drotrecogin Cohort vs Control Cohort; Test type: Superiority or Other; p = 0.871, Repeated Measures - propensity adjusted — 24-Hour Change from Baseline p-value

4. Secondary Outcome: Cardiovascular Performance Measures Obtained With a Pulmonary Artery Catheter - Cardiac Index
Description: Cardiac Index = cardiac output divided by body surface area.
Time Frame: Baseline to 24 Hours
Population: Number of per-protocol participants with values at baseline and 24 hours.
Measure: Mean (Standard Deviation); unit: liters/minute/meters squared
Arm/Group | Drotrecogin Cohort | Control Cohort
Number analyzed (Participants) | 17 | 13
liters/minute/meters squared
  24 Hours | 3.3 (0.7) | 3.2 (1.0)
  24 Hour Change from Baseline | -0.2 (1.5) | 0.1 (0.9)
Statistical Analysis 1: Comparison: Drotrecogin Cohort vs Control Cohort; Test type: Superiority or Other; p = 0.704, Repeated Measures - propensity adjusted — 24-Hour p-value
Statistical Analysis 2: Comparison: Drotrecogin Cohort vs Control Cohort; Test type: Superiority or Other; p = 0.702, Repeated Measures - propensity adjusted — 24-Hour Change from Baseline p-value

5. Secondary Outcome: Lactate Level
Description: Measures of global tissue perfusion and oxygenation were assessed via lactate levels.
Time Frame: Baseline to 6 Hours
Population: Number of per-protocol participants with values at baseline and 6 hours.
Measure: Mean (Standard Deviation); unit: millimoles per Liter
Arm/Group | Drotrecogin Cohort | Control Cohort
Number analyzed (Participants) | 19 | 15
millimoles per Liter
  6 Hours | 1.8 (1.0) | 2.8 (4.6)
  6 Hour Change from Baseline | -0.2 (0.6) | 0.4 (1.7)
Statistical Analysis 1: Comparison: Drotrecogin Cohort vs Control Cohort; Test type: Superiority or Other; p = 0.061, Repeated Measures - propensity adjusted — 6-Hour p-value
Statistical Analysis 2: Comparison: Drotrecogin Cohort vs Control Cohort; Test type: Superiority or Other; p = 0.027, Repeated Measures - propensity adjusted — 6-Hour Change from Baseline p-value

6. Secondary Outcome: Microcirculatory Measures From Sidestream Darkfield (SDF) Microscopy - Small Vessel Microvascular Flow Index (MFI)
Description: Per vessel category (and per quadrant), scored flow as follows: no flow=0, intermediate flow=1, sluggish flow=2, continuous flow=3. The MFI per vessel category calculated with formula (Q1+Q2+Q3+Q4)/4. Scores could range from 0 (sluggish flow) to 3 (continuous flow).
Time Frame: Baseline to 24 Hours
Population: Number of per-protocol participants with values at baseline, 12, and 24 hours.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Drotrecogin Cohort | Control Cohort
Number analyzed (Participants) | 19 | 18
units on a scale
  Baseline | 2.70 (0.51) | 2.50 (0.70)
  12 Hour | 2.95 (0.13) | 2.80 (0.35)
  24 Hour | 2.56 (0.83) | 2.65 (0.47)
  24 Hour Change from Baseline | -0.21 (0.61) | 0.06 (0.27)
Statistical Analysis 1: Comparison: Drotrecogin Cohort vs Control Cohort; Test type: Superiority or Other; p = 0.242, Repeated Measures - propensity adjusted — Baseline p-value
Statistical Analysis 2: Comparison: Drotrecogin Cohort vs Control Cohort; Test type: Superiority or Other; p = 0.083, Repeated Measures - propensity adjusted — 12-Hour p-value
Statistical Analysis 3: Comparison: Drotrecogin Cohort vs Control Cohort; Test type: Superiority or Other; p = 0.810, Repeated Measures - propensity adjusted — 24-Hour p-value
Statistical Analysis 4: Comparison: Drotrecogin Cohort vs Control Cohort; Test type: Superiority or Other; p = 0.623, Repeated Measures - propensity adjusted — 24-Hour Change from Baseline p-value

7. Secondary Outcome: Sequential Organ Failure Assessment (SOFA) Score at Baseline and 24 Hours
Description: The presence of 5 organ dysfunctions (cardiovascular, respiratory, renal, hepatic, coagulation) was assessed using a Sequential Organ Failure Assessment (SOFA) score. Each organ has a possible dysfunction score of 0 to 4, for a total SOFA score range of 0 (no organ dysfunction) to 20 (all organs with dysfunction).
Time Frame: Baseline and 24 Hours
Population: Number of per-protocol participants with values at baseline and 24 hours.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Drotrecogin Cohort | Control Cohort
Number analyzed (Participants) | 19 | 19
units on a scale
  Baseline | 8.5 (2.0) | 8.3 (3.2)
  24 Hours | 7.8 (2.3) | 7.8 (4.0)
Statistical Analysis 1: Comparison: Drotrecogin Cohort vs Control Cohort; Test type: Superiority or Other; p = 0.686, Repeated Measures - propensity adjusted — Baseline p-value
Statistical Analysis 2: Comparison: Drotrecogin Cohort vs Control Cohort; Test type: Superiority or Other; p = 0.575, Repeated Measures - propensity adjusted — 24-Hour p-value

8. Secondary Outcome: Change From Baseline in Creatinine Clearance (CrCl) at 24 Hours
Description: CrCl = (urine creatinine*urine volume)/(plasma creatinine*time period of urine collection). Corrected CrCl = CrCl*1.73/body surface area. Change in CrCl = Endpoint minus baseline.
Time Frame: Baseline and 24 hours
Population: Number of per-protocol participants with values at baseline and 24 hours.
Measure: Mean (Standard Deviation); unit: milliliter per minute
Arm/Group | Drotrecogin Cohort | Control Cohort
Number analyzed (Participants) | 15 | 8
milliliter per minute | -9.74 (75.45) | 1.66 (28.90)
Statistical Analysis 1: Comparison: Drotrecogin Cohort vs Control Cohort; Test type: Superiority or Other; p = 0.165, Repeated Measures - propensity adjusted

9. Secondary Outcome: 7 Day All-cause In-hospital Mortality
Time Frame: baseline to 7 days
Population: All enrolled patients
Measure: Number; unit: partipants
Arm/Group | Drotrecogin Cohort | Control Cohort
Number analyzed (Participants) | 22 | 21
partipants
  Alive at 7 Days | 18 | 13
  Not Alive at 7 Days | 4 | 8

10. Secondary Outcome: Endogenous Protein C Level
Time Frame: Baseline to 24 Hours
Population: Number of per-protocol participants with values at baseline, 12, and 24 hours.
Measure: Mean (Standard Deviation); unit: percentage of Protein C activity
Arm/Group | Drotrecogin Cohort | Control Cohort
Number analyzed (Participants) | 16 | 18
percentage of Protein C activity
  Baseline | 38.7 (25.2) | 34.8 (19.1)
  12 Hours | 48.2 (23.0) | 38.9 (19.6)
  24 Hours | 54.7 (20.7) | 40.0 (17.9)
  24 Hour Change from Baseline | 16.3 (16.2) | 2.4 (16.7)
Statistical Analysis 1: Comparison: Drotrecogin Cohort vs Control Cohort; Test type: Superiority or Other; p = 0.552, Repeated Measures - propensity adjusted — Baseline p-value
Statistical Analysis 2: Comparison: Drotrecogin Cohort vs Control Cohort; Test type: Superiority or Other; p = 0.129, Repeated Measures - propensity adjusted — 12-Hour p-value
Statistical Analysis 3: Comparison: Drotrecogin Cohort vs Control Cohort; Test type: Superiority or Other; p = 0.030, Repeated Measures - propensity adjusted — 24-Hour p-value
Statistical Analysis 4: Comparison: Drotrecogin Cohort vs Control Cohort; Test type: Superiority or Other; p = 0.002, Repeated Measures - propensity adjusted — 24-Hour Change from Baseline p-value

11. Other Pre Specified Outcome: Number of Participants With Bleeding Events
Description: Serious bleeding event resulted in one of following outcomes, or was significant for any reason: initial/ prolonged inpatient hospitalization; life-threatening experience; persistent or significant disability/incapacity; congenital anomaly/birth defect. Intracranial hemorrhage was also considered serious bleeding event.
Time Frame: baseline to 7 days
Population: All enrolled patients
Measure: Number; unit: participants
Arm/Group | Drotrecogin Cohort | Control Cohort
Number analyzed (Participants) | 22 | 21
participants
  Serious Bleeding Event | 2 | 0
  Intracranial Hemorrhage | 0 | 0

12. Secondary Outcome: Mixed Venous Oxygen Saturation
Description: Cardiovascular performance measures obtained with a pulmonary catheter as assessed by mixed venous oxygen saturation.
Time Frame: Baseline to 24 Hours
Population: Number of per-protocol participants with values at baseline and 24 hours.
Measure: Mean (Standard Deviation); unit: percent saturation mixed venous oxygen
Arm/Group | Drotrecogin Cohort | Control Cohort
Number analyzed (Participants) | 15 | 14
percent saturation mixed venous oxygen
  24 Hours | 69.6 (8.3) | 75.0 (11.1)
  24 Hour Change from Baseline | 3.7 (14.5) | 6.5 (13.3)
Statistical Analysis 1: Comparison: Drotrecogin Cohort vs Control Cohort; Test type: Superiority or Other; p = 0.128, Repeated Measures - propensity adjusted — 24-Hour p-value
Statistical Analysis 2: Comparison: Drotrecogin Cohort vs Control Cohort; Test type: Superiority or Other; p = 0.234, Repeated Measures - propensity adjusted — 24-Hour Change from Baseline p-value

ADVERSE EVENTS:
Arm/Group | Drotrecogin Cohort | Control Cohort
Serious Adverse Events (participants affected / at risk) | 4 | 3
Other Adverse Events (participants affected / at risk) | 4 | 0
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Drotrecogin Cohort | Control Cohort
Bradycardia (Cardiac disorders) | 0/22 (0) | 2/21 (2)
Cardiac arrest (Cardiac disorders) | 1/22 (1) | 0/21 (0)
Ventricular tachycardia (Cardiac disorders) | 1/22 (1) | 2/21 (2)
Right sided hemothorax (Injury, poisoning and procedural complications) | 1/22 (2) | 0/21 (0)
Hemorrage intraperitoneal (Vascular disorders) | 1/22 (1) | 0/21 (0)
OTHER ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Drotrecogin Cohort | Control Cohort
Atrial fibrilation (Cardiac disorders) | 1/22 (1) | 0/21 (0)
Gastrointestinal bleeding (Gastrointestinal disorders) | 1/22 (1) | 0/21 (0)
Gross hematuria (Renal and urinary disorders) | 1/22 (1) | 0/21 (0)
Oropharynx blood and ecchymoses (Skin and subcutaneous tissue disorders) | 1/22 (1) | 0/21 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days